CLINICAL TRIAL: NCT07363434
Title: RESONATE Study: Real-world Outcomes With Ribociclib in Indian Patients With HR+, HER2- Advanced Breast Cancer
Brief Title: A Real-world Study of Indian Patients With Advanced Breast Cancer Treated With Ribociclib
Acronym: RESONATE
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011AIN01
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Ribociclib; Endocrine therapy; Metastasis; Progression-free survival
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Ribociclib Group: Indian women with a confirmed diagnosis of HR+, HER2- aBC who were treated with ribociclib in combination with ET.

SUMMARY:
The aim of this study was to assess the effectiveness, safety, and tolerability of ribociclib in Indian women with hormone receptor positive (HR+) and human epidermal growth factor receptor 2 negative (HER2-) advanced breast cancer (aBC).

This study used secondary data sources, i.e., paper-based records; electronic medical records (EMRs); and other sources, such as radiology reports, pathology reports, and examination/clinician notes related to aBC, from clinics/hospitals across 18 sites in India. Aggregated data of anonymized patients treated with ribociclib plus endocrine therapy (ET) by the approved indication between June 2018 and December 2021 were collected and analyzed.

ELIGIBILITY:
Inclusion criteria:

• Women ≥18 years old diagnosed with HR+ and HER2- aBC who received at least one dose of ribociclib in combination with ET following the approved indication, with at least one follow-up visit after diagnosis or death due to any cause.

Exclusion criteria:

• Patients with prior/current enrollment in an interventional clinical trial for aBC/metastatic breast cancer and those who had received another cyclin-dependent kinase 4 and 6 (CDK4/6) inhibitor in any setting.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included HR+/HER2- aBC patients who received ribociclib in combination with ET in India.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Real-world Progression-free Survival (rwPFS) for the Entire Patient Group | Up to approximately 42 months
  rwPFS was defined as the time from the start of ribociclib treatment in combination with ET to disease progression, as assessed by the treating physician, or death due to any cause.
rwPFS by Line of Therapy for the Entire Patient Group | Up to approximately 42 months
  rwPFS was defined as the time from the start of ribociclib treatment in combination with ET to disease progression, as assessed by the treating physician, or death due to any cause.
Duration of Clinical Response by Type of Clinical Response and Line of Therapy for the Entire Patient Group | Up to approximately 42 months
  Clinical response categories included complete response, any response (other than complete response), no response, and any progression.
Number of Patients by Type of Clinical Response and Line of Therapy for the Entire Patient Group | Up to approximately 42 months
  Clinical response categories included complete response, any response (other than complete response), no response, and any progression.

SECONDARY OUTCOMES:
rwPFS for Patients With at Least 6 Months of Follow-up | Up to approximately 42 months
  rwPFS was defined as the time from the start of ribociclib treatment in combination with ET to disease progression, as assessed by the treating physician, or death due to any cause.
rwPFS by Line of Therapy for Patients With at Least 6 Months of Follow-up | Up to approximately 42 months
  rwPFS was defined as the time from the start of ribociclib treatment in combination with ET to disease progression, as assessed by the treating physician, or death due to any cause.
Duration of Clinical Response by Type of Clinical Response and Line of Therapy for Patients With at Least 6 Months of Follow-up | Up to approximately 42 months
  Clinical response categories included complete response, any response (other than complete response), no response, and any progression.
Number of Patients With Adverse Events | Up to approximately 42 months
Number of Adverse Events | Up to approximately 42 months
Number of Adverse Events by Severity | Up to approximately 42 months
Number of Patients who Discontinued Treatment by Reason for Discontinuation | Up to approximately 42 months
Number of Patients by Adverse Event That Led to Dose Discontinuation | Up to approximately 42 months
Number of Patients by Adverse Event That Led to Dose Interruptions | Up to approximately 42 months
Number of Patients by Adverse Event That Led to Dose Reduction | Up to approximately 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States